CLINICAL TRIAL: NCT04794556
Title: Respiratory Protection Effect of Ear-loop-type KF94 Filtering Facepiece Respirators According to the Wearing Method: A Randomized, Open-label Study
Brief Title: Respiratory Protection Effect of Ear-loop-type KF94 Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hee Yoon, Clinical Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KF94 mask
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Infection
Keywords: Respiratory protective devices; quantitative fit test; N95 filtering facepiece respirators; infection control; KF94 mask
MeSH Terms: conditions — Infections | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants were randomly assigned to groups A, B, and C to reduce learning effects according to the mask type
  Interventions: Device: tight-fitting of KF94 mask with clip
- Group B (Experimental): Participants were randomly assigned to groups A, B, and C to reduce learning effects according to the mask type
  Interventions: Device: tight-fitting of KF94 mask with clip
- Group C (Experimental): Participants were randomly assigned to groups A, B, and C to reduce learning effects according to the mask type
  Interventions: Device: tight-fitting of KF94 mask with clip

INTERVENTIONS:
Device: tight-fitting of KF94 mask with clip — The general-fitting method involved wearing a mask with ear loops, and the tight-fitting method involved wearing a clip that connected ear loops on the occiput after wearing a mask according to the general method

SUMMARY:
Ear-loop-type Korean Filter 94 masks (KF94 masks, equivalent to the N95 and FFP2) are broadly used in health care settings in Korea for the COVID-19 pandemic. However, no studies have assessed the adequacy of respiratory protection. In this prospective randomized open-label study, the investigators aimed to evaluate the fitting performance of ear-loop-type KF94 masks by the quantitative fit test according to the occupational safety and health administration (OSHA) protocol. In addition, by quantitatively comparing the "tight-fitting" method using a clip and the "general-fitting" method, the investigators tried to evaluate whether the tight-wearing method improves the fitting performance of KF94 masks.

DETAILED DESCRIPTION:
Sample size: The sample size was calculated based on a pilot study of 10 participants, which examined the FF of general-fitting. The mean FF was 20.3, and the log-transformed FFs were assessed due to skewed data, which was 1.98 (standard deviation 1.34). We assumed that the FF for tight-fitting would increase by 50%, with an α value of .05, and a β error of .10 (power = 90%) for two-sided hypothesis testing. The estimated sample size calculation revealed a required sample of 24 participants. Therefore, 30 participants were enrolled to account for a 20% dropout rate.

Data analyses: Repeated-measures analysis of variance or generalized estimating equations were used to compare the FFs or passing rate of the QNFTs for the three mask types according to the wearing method. Paired t-tests or Wilcoxon signed-rank tests were used to compare the FFs according to the wearing method for each mask type. McNemar's test was used to compare the passing rate of the QNFT according to the wearing method. Bonferroni's correction was performed for all results of each subgroup analysis. SAS ver. 9.4 software (SAS Institute, Cary, NC) was used to perform all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* healthcare workers with experience in wearing filtering facepiece respirator working in the hospital

Exclusion Criteria:

* Individuals with expected difficulties in wearing masks or undergoing OSHA fit tests because of factors such as a facial anomaly, lung disease, or lower back disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
total fit factors(FFs) of the quantitative fit tests (QNFT) according to the wearing method of the three types of KF94 masks | through study completion, an average of 1 year

SECONDARY OUTCOMES:
passing rate of the QNFT according to the wearing method | through study completion, an average of 1 year
total FFs after user-seal-check and real-time adjustment | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yoon, MD., PhD., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang HJ, Yoon H, Kang SY, Lee G, Park JE, Kim T, Lee SU, Hwang SY, Cha WC, Shin TG, Jo IJ. Respiratory Protection Effect of Ear-loop-type KF94 Masks according to the Wearing Method in COVID-19 Pandemic: a Randomized, Open-label Study. J Korean Med Sci. 2021 Jul 19;36(28):e209. doi: 10.3346/jkms.2021.36.e209. PMID 34282608